CLINICAL TRIAL: NCT07184502
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single and Multiple Ascending Dose Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ZT003 Injection in Healthy Volunteers and Overweight or Obese Volunteers
Brief Title: Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of ZT003 Injection Following Single and Multiple Subcutaneous Administration in Healthy Volunteers/Overweight or Obese Volunteers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing QL Biopharmaceutical Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BJQL-ZT003-1001
Record Dates: First submitted 2025-08-19; First posted 2025-09-22 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Up to 5 Single Ascending Dose (SAD) Cohorts - ZT003 (Experimental): Participants will receive a single subcutaneous dose of ZT003 at ascending dose levels across up to 5 cohorts.
  Interventions: Drug: ZT003
- Up to 3 Multiple Ascending Dose (MAD) Cohorts - ZT003 (Experimental): Participants will receive multiple subcutaneous doses of ZT003 at ascending dose levels across up to 3 cohorts.
  Interventions: Drug: ZT003
- SAD/MAD Placebo (Placebo Comparator): Participants will receive either a single or multiple subcutaneous doses of placebo, corresponding to the dosing schedule of the respective cohort (SAD or MAD).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ZT003 — ZT003 is administered as a single subcutaneous injection at different dose levels.
  Arms: Up to 5 Single Ascending Dose (SAD) Cohorts - ZT003
Drug: ZT003 — ZT003 administered as multiple subcutaneous injections at different dose levels.
  Arms: Up to 3 Multiple Ascending Dose (MAD) Cohorts - ZT003
Drug: Placebo — Matching placebo administered subcutaneously.
  Arms: SAD/MAD Placebo

SUMMARY:
This is a Phase 1, randomized, double-blind, placebo-controlled, single-center study designed to evaluate the safety, tolerability, and pharmacokinetics of ZT003 following subcutaneous administration in healthy adult participants. The study includes both single ascending dose (SAD) and multiple ascending dose (MAD) parts.

DETAILED DESCRIPTION:
This is a first-in-human, Phase 1, randomized, single-center, double-blind, placebo-controlled study to evaluate the safety, tolerability, and pharmacokinetics of ZT003 following subcutaneous administration in healthy adult participants. The study is designed in two parts:

Part A (Single Ascending Dose [SAD]): Approximately 40 participants will be enrolled into sequential dose cohorts. Each cohort will receive a single dose of ZT003 or matching placebo administered subcutaneously. Dose escalation will proceed based on safety, tolerability, and pharmacokinetic data from the preceding cohorts.

Part B (Multiple Ascending Dose [MAD]): Approximately 36 participants will be enrolled into sequential cohorts. Each participant will receive multiple subcutaneous doses of ZT003 or placebo. Dosing frequency and duration will be based on data obtained from Part A and guided by predefined criteria.

The study will evaluate safety through the monitoring of adverse events, clinical laboratory tests, vital signs, physical examinations, ECGs, and injection site assessments. Pharmacokinetic parameters will be measured using plasma drug concentration profiles. The results from this study will inform dose selection and design for future clinical studies in patient populations.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female participants, aged 18 to 65 years at the time of screening.
2. Body weight >50 kg to <130 kg, and BMI between 22.0 and 45.0 kg/m square.
3. Medically healthy, with no clinically significant abnormalities in medical history, physical examination, vital signs, ECG, or clinical laboratory assessments, as judged by the Investigator.
4. Females of childbearing potential must use highly effective contraception and have a negative pregnancy test at screening and Day -1.
5. Male participants must agree to use acceptable contraception from screening through at least 90 days after the last dose.
6. Able to understand and comply with study procedures and provide written informed consent.
7. Thyroid function tests within normal range as specified by the testing laboratory, unless deemed not clinically significant by the PI or designee.

Exclusion Criteria:

1. History or presence of any clinically significant disease or disorder that may put the participant at risk or interfere with study assessments.
2. Positive test for hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV Ab), or HIV antibody at screening.
3. History of drug or alcohol abuse within 12 months prior to screening.
4. Use of prescription drugs, over-the-counter medications, herbal products, or supplements within 14 days (or 5 half-lives) prior to first dose unless deemed acceptable by the Investigator.
5. Participation in another clinical study with an investigational product within 30 days or 5 half-lives of the investigational product before dosing.
6. Any history of significant allergy or hypersensitivity to any component of the investigational medicinal product (IMP).
7. Clinically significant ECG abnormalities, including QTc >450 ms (males) or >470 ms (females) at screening.
8. Abnormal clinical laboratory results at screening considered clinically significant by the Investigator.
9. History of bleeding disorders or current use of anticoagulant therapy.
10. Pregnant or lactating females, or females planning to become pregnant during the study period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-10-16 (Actual); Primary Completion 2026-06-06 (Estimated); Study Completion 2026-10-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAEs) | Collected at every visit (Screening, Day -1, Day 1 pre- and post-dose, Days 2-7, and follow-ups at Days 8, 15, 22, 29, and 36).
Incidence of Serious Adverse Events (SAEs) | Collected at every visit (Screening, Day -1, Day 1 pre- and post-dose, Days 2-7, and follow-ups at Days 8, 15, 22, 29, and 36).
Incidence of Adverse Events of Special Interest (AESIs) | Collected at every visit (Screening, Day -1, Day 1 pre- and post-dose, Days 2-7, and follow-ups at Days 8, 15, 22, 29, and 36).
Incidence of Adverse Events Leading to Study Drug Discontinuation or Withdrawal | Collected at every visit (Screening, Day -1, Day 1 pre- and post-dose, Days 2-7, and follow-ups at Days 8, 15, 22, 29, and 36).
Incidence and Severity of Injection Site Reactions (ISRs) | From first dose (Day 1) through End of Treatment/EOT visit (Day 85)
Change from Baseline in Systolic Blood Pressure | From Screening (Day -35) through End of Treatment (Day 85).
Change from Baseline in Diastolic Blood Pressure | From Screening (Day -35) through End of Treatment (Day 85).
Change from Baseline in Pulse Rate | From Screening (Day -35) through End of Treatment (Day 85).
Change from Baseline in Body Temperature | From Screening (Day -35) through End of Treatment (Day 85).
Change from Baseline in Respiratory Rate | From Screening (Day -35) through End of Treatment (Day 85).
Change from Baseline in ECG Heart Rate | From Screening (Day -35) through End of Treatment (Day 85).
Change from Baseline in ECG PR Interval | From Screening (Day -35) through End of Treatment (Day 85).
Change from Baseline in ECG QRS Duration | From Screening (Day -35) through End of Treatment (Day 85).
Change from Baseline in ECG QT Interval | From Screening (Day -35) through End of Treatment (Day 85).
Change from Baseline in ECG Corrected QT Interval (QTcF) | From Screening (Day -35) through End of Treatment (Day 85).

SECONDARY OUTCOMES:
Plasma Cmax of ZT003 | Day 1 to 24 hours post-dose (SAD); pre-dose to 24 hours post-final dose (MAD)
Plasma Tmax of ZT003 | Day 1 to 24 hours post-dose (SAD); pre-dose to 24 hours post-final dose (MAD)
AUC from time zero to the last quantifiable concentration of ZT003 | SAD: Day 1 to 96 hours post-dose; MAD: Pre-dose on Days 1, 8, 15, 22, and 29 to 96 hours post-final dose (Day 29), with additional samples up to Day 78 and at End of Treatment (Day 85).
AUC from time zero extrapolated to infinity of ZT003 | SAD: Day 1 to 96 hours post-dose; MAD: Pre-dose on Days 1, 8, 15, 22, and 29 to 96 hours post-final dose (Day 29), with additional samples up to Day 78 and at End of Treatment (Day 85).
Plasma half-life (t½) of ZT003 | SAD: Day 1 to 96 hours post-dose; MAD: Pre-dose on Days 1, 8, 15, 22, and 29 to 96 hours post-final dose (Day 29), with additional samples up to Day 78 and at End of Treatment (Day 85).
Apparent Clearance (CL/F) of ZT003 | SAD: Day 1 to 96 hours post-dose; MAD: Pre-dose on Days 1, 8, 15, 22, and 29 to 96 hours post-final dose (Day 29), with additional samples up to Day 78 and at End of Treatment (Day 85).
Apparent Volume of Distribution (Vz/F) of ZT003 | SAD: Day 1 to 96 hours post-dose; MAD: Pre-dose on Days 1, 8, 15, 22, and 29 to 96 hours post-final dose (Day 29), with additional samples up to Day 78 and at End of Treatment (Day 85).
Presence of Anti-Drug Antibodies (ADA) | Baseline, Day 29, Day 57, and End of Study (Day 85)

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network Brisbane, Brisbane, Queensland, Australia